CLINICAL TRIAL: NCT06669988
Title: Comparison of the Teaching Effectiveness of VR, Videos, and Written Materials on Food Hygiene Safety and Equipment Operation
Brief Title: Comparison of Teaching Effectiveness of VR, Video, and Written Materials on Food Hygiene and Equipment Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, SHIH, HSIN-YU, Principal Investigator, Fu Jen Catholic University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C112203
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Educational Interventions; Virtual Reality
Keywords: Virtual Reality; education; hygiene safety in food service

STUDY DESIGN:
Intervention Model Description: This study will include students from both nutrition and non-nutrition departments. Participants will engage in one of three teaching modes: VR group, video group, or written materials group, all focusing on hygiene safety during food service and equipment operation. In the VR group, participants will wear virtual reality headsets for immersive learning in a 3D space with interactive scenarios, simulating a large-scale food service environment. In the video group, participants will watch a 2D video featuring similar scenarios to the VR experience but without interactive elements. The written materials group will receive content through static photos and text, lacking dynamic visuals or immersive experiences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VR Group (Experimental): In the VR group, participants will wear virtual reality headsets, experiencing immersive learning in a 3D space with interactive scenarios. Interactive buttons will assist them, making it feel as if they are physically entering a large-scale food service environment. The immersive learning focuses on operating large kitchen equipment, and the first-person perspective will make participants feel as if they are truly in the environment, preparing food in real-time. The VR experience will cover everything from clothing regulations, hygiene and safety precautions, and the use of large kitchen equipment to food service procedures and emergency response. All these aspects are integrated into the learning process.
  Interventions: Device: VR
- Video Group (Experimental): In the video group, participants will watch a video that features scenarios similar to those in the VR experience. However, instead of interacting with a 3D space, the content will be presented in a 2D format without the immersive spatial element.
  Interventions: Device: Video
- Written Materials Group (Sham Comparator): In the written materials group, the content will be presented through photos and text, without offering dynamic visuals or the immersive 3D spatial experience.
  Interventions: Device: written materials

INTERVENTIONS:
Device: VR — VR - Immersive instruction using virtual reality.
  Arms: VR Group
Device: Video — Video - Educational content presented through video.
  Arms: Video Group
Device: written materials — Written Materials - Instruction using text and images.
  Arms: Written Materials Group

SUMMARY:
This study investigates the impact of virtual reality (VR) as an educational tool in the food industry, comparing it to traditional methods like videos and written materials in teaching hygiene and safety. VR offers immersive, realistic training that allows employees to simulate food-handling scenarios, including handwashing, hazard identification, and emergency responses, which may enhance engagement and effectiveness. The study aims to clarify the advantages and limitations of VR-based education against traditional approaches by assessing learning effectiveness, usefulness, playfulness, ease of use, and long-term knowledge retention.

Participants will be assigned to one of the three educational methods (VR, video, or written materials) and evaluated through pre-tests, post-tests, and follow-up assessments one month later. Non-parametric statistical analysis, specifically the Wilcoxon signed-rank test, will assess the effectiveness of each educational method based on test scores and satisfaction surveys.

The study will be conducted at Fu Jen Catholic University's Department of Nutrition, following ethical guidelines and informed consent protocols to protect participants' welfare and data privacy. Professional supervision and carefully maintained equipment will ensure a safe learning environment, with adverse reactions monitored and documented throughout.

DETAILED DESCRIPTION:
Virtual Reality (VR) is a rapidly evolving field with immense potential in education. In recent years, aside from medical education, VR is also growing in the food industry. Using VR, employees can receive realistic, immersive training experiences, enabling them to learn knowledge in hygiene and safety. The purpose of this shift in educational methods is to enhance the effectiveness of training for professionals. By using VR, employees can simulate real-life scenarios in restaurant, including tasks such as handling ingredients, practicing proper handwashing procedures, identifying and resolving potential hazards, and responding to emergency situations. VR in hygiene and safety education offers numerous benefits to the food industry. Therefore, this study aims to explore whether VR can replace or complement traditional educational methods in original course. By using different educational methods, including VR, videos, and written materials, the study seeks to clarify the advantages and disadvantages of traditional education and technology-based education. Building on the original course, this study compares the learning effectiveness, usefulness, playfulness, ease of use, and long-term knowledge retention of these three educational methods.

The statistical method planned for this study is non-parametric analysis, specifically the Wilcoxon signed-rank test, to analyze the participants' data. The evaluation of results will focus on the learning effectiveness assessment, with the primary evaluation indicators being the scores from the pre-test, post-test, and VR post-test. One month later, a re-evaluation of knowledge retention will be conducted. In the satisfaction survey, the main aspects assessed will be usefulness, playfulness, ease of use.

This study will first use a written consent form to ensure that participants fully understand the study's purpose, procedures, potential risks, and benefits. The consent form will include the following key information: the purpose of the study, the research procedures and possible risks, privacy protection measures for participants, voluntary participation, and the right to withdraw from the study at any time.

The researchers will explain the study plan in detail to the participants during the initial meeting and answer any questions they may have. This activity will take place in a classroom at Fu Jen Catholic University's Department of Nutrition. Participants will have sufficient time to read and understand the consent form thoroughly, and they will be able to ask questions before signing it. There will be two copies of the consent form: one for the participant to keep and another for the research team to archive, ensuring the safety and protection of participants. This study will ensure that all instructional activities are conducted under professional supervision, using well-tested and properly maintained equipment. While using the VR equipment, participants will be guided by trained professionals to avoid any discomfort or injuries that may result from improper use. If participants experience any adverse reactions during the study, such as dizziness, eye fatigue, or emotional discomfort, their participation will be immediately halted, and on-site personnel will provide an initial assessment and appropriate care. All adverse events will be documented and reported to the study principal investigator. If necessary, further evaluations will be conducted to determine if adjustments to the study protocol or procedures are required.

This study will strictly adhere to personal data protection regulations to ensure the confidentiality and security of all participants' information. Participants' identities will not be disclosed in any research reports or publications. These measures will help ensure that the study complies with ethical guidelines, respects the rights and welfare of participants, and addresses any potential adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* native Chinese speakers
* normal vision, hearing, and hand mobility

Exclusion Criteria:

* in other VR-related studies
* symptoms of dizziness when wearing a virtual reality headset
* have taken courses in food service or food hygiene and safety

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
learning effectiveness assessment | an hour
  Primary evaluation indicators being the scores from the pre-test, post-test, and VR post-test.
knowledge retention | From enrollment to one month after the completion of the teaching intervention.
  Re-evaluation indicators being the scores from the post-test, and VR post-test.
user experience feedback | an hour
  A total of 12 questions, using a satisfaction rating scale from 1 to 5, with 5 being the highest score. The main content includes ease of use of the VR equipment, whether it enhances learning motivation, understanding of spatial concepts, and skills in food service.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksoy E. Comparing the Effects on Learning Outcomes of Tablet-Based and Virtual Reality-Based Serious Gaming Modules for Basic Life Support Training: Randomized Trial. JMIR Serious Games. 2019 May 1;7(2):e13442. doi: 10.2196/13442. PMID 31042153
- [Background] Chao YC, Hu SH, Chiu HY, Huang PH, Tsai HT, Chuang YH. The effects of an immersive 3d interactive video program on improving student nurses' nursing skill competence: A randomized controlled trial study. Nurse Educ Today. 2021 Aug;103:104979. doi: 10.1016/j.nedt.2021.104979. Epub 2021 May 18. PMID 34049120
- [Background] Makinen H, Haavisto E, Havola S, Koivisto JM. Graduating nursing students' user experiences of the immersive virtual reality simulation in learning - A qualitative descriptive study. Nurs Open. 2023 May;10(5):3210-3219. doi: 10.1002/nop2.1571. Epub 2023 Jan 4. PMID 36598872
- See also: Kwon, C. Verification of the possibility and effectiveness of experiential learning using HMD-based immersive VR technologies. Virtual Reality 2019; 23: 101-118. — https://doi.org/10.1007/s10055-018-0364-1
- See also: Karanezi, X., E. Rapti, and G. Halimi Traditional and Modern Teaching Methodologies: Which One is More Successful and What are the Challenges? Academic Journal of Interdisciplinary Studies 2015; 4: 311. — https://doi.org/10.5901/ajis.2015.v4n2s2p311
- See also: Pan, Z., et al. Virtual reality and mixed reality for virtual learning environments. Computers & Graphics 2006; 30: 20-28. — https://doi.org/10.1016/j.cag.2005.10.004
- See also: Clark, J., P. Crandall, and J. Shabatura Wearable Technology Effects on Training Outcomes of Restaurant Food Handlers. Journal of Food Protection 2018; 81: 1220-1226. — https://doi.org/10.4315/0362-028X.JFP-18-033
- See also: Mikropoulos, T.A. and A. Natsis Educational virtual environments: A ten-year review of empirical research (1999-2009). Computers & Education 2011; 56: 769-780. — https://doi.org/10.1016/j.compedu.2010.10.020
- See also: Merchant, Z., et al. Effectiveness of virtual reality-based instruction on students' learning outcomes in K-12 and higher education: A meta-analysis. Computers & Education 2014; 70: 29-40. — https://doi.org/10.1016/j.compedu.2013.07.033